CLINICAL TRIAL: NCT05902117
Title: Place of Copeptin-troponin Assay in the Elimination Diagnosis of Non-ST+ ACS in the Management of Pre-hospital and In-hospital Non-traumatic Chest Pain in Adults
Brief Title: Place of Copeptin-troponin Assay in the Elimination Diagnosis of Non-ST+ ACS
Acronym: CopSCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHRD0821
Record Dates: First submitted 2023-05-11; First posted 2023-06-13 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-06

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction; Troponine; Copeptine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Troponin and Copeptin assay (Experimental): Collection of an additional blood tube for copeptin determination during blood collection for troponin testing as part of care.
  Interventions: Diagnostic Test: Troponin and Copeptin assay

INTERVENTIONS:
Diagnostic Test: Troponin and Copeptin assay — Collection of an additional blood tube for copeptin determination during blood collection for troponin testing as part of care.

SUMMARY:
The aim of this study is to demonstrate that a combined troponin and copeptin assay can exclude non-ST+ ACS in patients with chest pain less than 6 hours old.

DETAILED DESCRIPTION:
Chest pain accounts for about 10% of emergency service visits, which represents between 6 and 8 million visits per year in the United States and 15 million in Europe. Depending on the series, coronary etiology is found in 10 to 50% of cases.

Two types of coronary syndrome are distinguished according to the existence of a pathological change in the electrocardiogram.

ST+ acute coronary syndrome is a diagnosis based on the association of chest pain associated with an electrocardiogram change in the form of ST-segment elevation in a systemic territory corresponding to the complete obstruction of an artery of the coronary network.

Non-ST+ coronary syndrome is more difficult to diagnose, as the ECG is not pathological or cannot be interpreted due to the presence of conduction disorders. The diagnosis is currently based on the pathological increase of a specific myocardial biomarker in the blood: troponin.

If the pain is recent (less than six hours) the troponin measured on arrival may be falsely negative, and therefore requires a second measurement 3 hours after the first one (this is the troponin cycle). This second test therefore leads to a longer stay for patients requiring it and contributes to the saturation of the emergency service.

Copeptin is an endogenous stress biomarker that rises immediately during a myocardial infarction and decreases rapidly. Unlike troponin, this marker is not myocardial specific and its level can rise in the blood for many reasons, which is why this marker cannot be used alone in the diagnosis of non-ST+ acute coronary syndrome (non-ST+ ACS or ST- ACS).

The hypothesis would be that the association of a copeptin assay with the initial troponin assay could, if both markers are below pathological thresholds (Troponin < 16ng.dL), eliminate the diagnosis of acute coronary syndrome from the first assays and thus avoid the second troponin assay 3 hours after the first. The patient would reduce the time spent in the emergency and would thus reduce the number of patients in the emergency service.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥18 years old
* Presenting at the Pontoise emergency department by their own means / ambulance or patients taken care of by the SMUR and referred to the NOVO hospital - Pontoise site
* Chest pain less than 6 hours old
* Chest pain suggestive of ACS (compressive, intense pain, radiating into the arm and neck, mid-thoracic, left thoracic or epigastric location)
* Non-contributory ECG (no ST elevation, presence of bundle branch block)
* Informed and having expressed no objection
* Beneficiary of a social security system (or entitled person)

Non -Inclusion Criteria:

* Sus ST-segment shift on ECG (ACS ST+)
* Intermittent pain/unclear onset time
* Pregnant woman
* Pain in the context of trauma
* Patient under guardianship
* Patient does not speak or understand French

Exclusion Criteria:

* Non-ultrasensitive troponin measurement positive during the 1st SMUR sampling (> 0.08 ng.dL)
* Patient not referred to the NOVO hospital - Pontoise site by the SMUR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Demonstrate that a combined troponin and copeptin assay can exclude non-ST+ ACS in patients with chest pain less than 6 hours old (sensitivity/specificity) | At the end of the study, an average of 8 month
  Comparison of copeptin and troponin assays in the final diagnosis of non-ST+ ACS based on emergency medical records by calculation the sensitivity/specificity of the troponin - copeptin pair.
Demonstrate that a combined troponin and copeptin assay can exclude non-ST+ ACS in patients with chest pain less than 6 hours old (negative predictive value) | At the end of the study, an average of 8 month
  Comparison of copeptin and troponin assays in the final diagnosis of non-ST+ ACS based on emergency medical records by calculation of the negative predictive value of the troponin - copeptin pair.

SECONDARY OUTCOMES:
Evaluation of the diagnostic performance (sensitivity/specificity) of the troponin/ copeptin association according to cardiovascular risk factors (age, smoking, hypertension, history of cardiac ischemia, overweight, heredity) | At the end of the study, an average of 8 month
  Evaluation of the diagnostic performance (sensitivity/specificity) of the troponin - copeptin pair for each subgroup of cardiovascular risk factors (age / smoking / hypertension / history of cardiac ischemia / overweight and heredity).
Evaluation of the diagnostic performance (negative predictive value) of the troponin/ copeptin association according to cardiovascular risk factors (age, smoking, hypertension, history of cardiac ischemia, overweight, heredity) | At the end of the study, an average of 8 month
  Evaluation of the diagnostic performance (negative predictive value) of the troponin - copeptin pair for each subgroup of cardiovascular risk factors (age / smoking / hypertension / history of cardiac ischemia / overweight and heredity).
Evaluation of the patient's length of stay | At the end of the Study, an average of 8 month
  Collection of the number of days or hours spent in the emergency service from the time of arrival
Evaluation of the diagnostic performance of the troponin/ copeptin combination according to the time from onset of pain | At the end of the study, an average of 8 month
  The diagnostic performance of the troponin/ copeptin combination is evaluated according to the time between the first pain and blood sampling
Evaluation of pain management in emergency service | At the end of the study, an average of 8 month
  Assessment of the evolution of pain via the numerical scale (EN), rated from 0 to 10, between arrival in the emergency room and reassessment at 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dr Olivier Fancelli, Principal Investigator — NOVO Hospital - Pontoise Site
Locations (2):
- France (2):
  - Emergency Department (SAMU) Hospital NOVO - Pontoise site, Pontoise
  - Emergency Service - UHCD Hospital NOVO - Pontoise site, Pontoise

REFERENCES:
- [Background] Mockel M, Searle J, Muller R, Slagman A, Storchmann H, Oestereich P, Wyrwich W, Ale-Abaei A, Vollert JO, Koch M, Somasundaram R. Chief complaints in medical emergencies: do they relate to underlying disease and outcome? The Charite Emergency Medicine Study (CHARITEM). Eur J Emerg Med. 2013 Apr;20(2):103-8. doi: 10.1097/MEJ.0b013e328351e609. PMID 22387754
- [Background] Fanaroff AC, Rymer JA, Goldstein SA, Simel DL, Newby LK. Does This Patient With Chest Pain Have Acute Coronary Syndrome?: The Rational Clinical Examination Systematic Review. JAMA. 2015 Nov 10;314(18):1955-65. doi: 10.1001/jama.2015.12735. PMID 26547467
- [Background] Dawson C, Benger JR, Bayly G. Serial high-sensitivity troponin measurements for the rapid exclusion of acute myocardial infarction in low-risk patients. Emerg Med J. 2013 Jul;30(7):593-4. doi: 10.1136/emermed-2012-201574. Epub 2012 Jul 31. PMID 22851671
- [Background] Khan SQ, Dhillon OS, O'Brien RJ, Struck J, Quinn PA, Morgenthaler NG, Squire IB, Davies JE, Bergmann A, Ng LL. C-terminal provasopressin (copeptin) as a novel and prognostic marker in acute myocardial infarction: Leicester Acute Myocardial Infarction Peptide (LAMP) study. Circulation. 2007 Apr 24;115(16):2103-10. doi: 10.1161/CIRCULATIONAHA.106.685503. Epub 2007 Apr 9. PMID 17420344
- [Background] Kim KS, Suh GJ, Song SH, Jung YS, Kim T, Shin SM, Kang MW, Lee MS. Copeptin with high-sensitivity troponin at presentation is not inferior to serial troponin measurements for ruling out acute myocardial infarction. Clin Exp Emerg Med. 2020 Mar;7(1):35-42. doi: 10.15441/ceem.19.013. Epub 2020 Mar 31. PMID 32252132
- [Background] Szarpak L, Lapinski M, Gasecka A, Pruc M, Drela WL, Koda M, Denegri A, Peacock FW, Jaguszewski MJ, Filipiak KJ. Performance of Copeptin for Early Diagnosis of Acute Coronary Syndromes: A Systematic Review and Meta-Analysis of 14,139 Patients. J Cardiovasc Dev Dis. 2021 Dec 27;9(1):6. doi: 10.3390/jcdd9010006. PMID 35050216
- [Background] Aarts GWA, van der Wulp K, Camaro C. Pre-hospital point-of-care troponin measurement: a clinical example of its additional value. Neth Heart J. 2020 Oct;28(10):514-519. doi: 10.1007/s12471-020-01434-w. PMID 32514934
- [Background] Kohn MA, Kwan E, Gupta M, Tabas JA. Prevalence of acute myocardial infarction and other serious diagnoses in patients presenting to an urban emergency department with chest pain. J Emerg Med. 2005 Nov;29(4):383-90. doi: 10.1016/j.jemermed.2005.04.010. PMID 16243193
- [Background] Charpentier S, Beaune S, Joly LM, Khoury A, Duchateau FX, Briot R, Renaud B, Ageron FX; IRU Network. Management of chest pain in the French emergency healthcare system: the prospective observational EPIDOULTHO study. Eur J Emerg Med. 2018 Dec;25(6):404-410. doi: 10.1097/MEJ.0000000000000481. PMID 28723703
- [Background] Hamm CW, Bassand JP, Agewall S, Bax J, Boersma E, Bueno H, Caso P, Dudek D, Gielen S, Huber K, Ohman M, Petrie MC, Sonntag F, Uva MS, Storey RF, Wijns W, Zahger D; ESC Committee for Practice Guidelines. ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: The Task Force for the management of acute coronary syndromes (ACS) in patients presenting without persistent ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2011 Dec;32(23):2999-3054. doi: 10.1093/eurheartj/ehr236. Epub 2011 Aug 26. No abstract available. PMID 21873419
- See also: Does This Patient With Chest Pain Have Acute Coronary Syndrome? — https://doi.org/10.1007/s13341-013-0370-6
- See also: Risk stratification of acute coronary syndromes (ST+ and non-ST+) — https://www.sfmu.org/upload/70_formation/02_eformation/02_congres/Urgences/urgences2012/donnees/pdf/013_charpentier.pdf